CLINICAL TRIAL: NCT01701245
Title: A Randomized, Multicenter Study for the Prevention and Acute Treatment of Chronic Cluster Headache Using Gammacore, Versus Standard of Care.
Brief Title: Prevention and Acute Treatment of Chronic Cluster Headache Compared to Standard of Care
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ElectroCore INC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC-002
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Results first posted 2016-04-25 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Cluster Headache
Keywords: vagus nerve stimulation; vagal nerve stimulation; nVNS; VNS; cluster headache; chronic; non invasive; gammacore
MeSH Terms: conditions — Cluster Headache; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of care (No Intervention): No intervention, standard of care
- GammaCore (Active Comparator): Three stimulation treatments 2x/day 7 to 10 hours apart from one another. In addition, three stimulation treatments at the time of onset of symptoms of a headache attack.
  Interventions: Device: GammaCore

INTERVENTIONS:
Device: GammaCore — vagal stimulation
  Arms: GammaCore

SUMMARY:
Subjects enrolled into this 10 week study will for the first two weeks document the number of cluster headaches and the means of treating (medication) of these attacks. Subjects will then be randomized to into either two groups. The first group is continuing with standard of care and the second group is treatment with the investigational device (GammaCore) for a period of 4 weeks. After this 4 week period, all subjects will treat with the GammaCore for another 4 week period. It is hypothesized the the treatment group will have a reduction in mean cluster headaches per week by 50% compared to the standard of care group.

DETAILED DESCRIPTION:
The study is a prospective randomized controlled multi-center investigation designed for comparison of two parallel groups, GammaCore® (active treatment) and Standard of Care, SoC, (control). The study period begins with a 2 week run-in period, followed by a 4 week comparative period when the subjects are randomized to either active treatment or control 1:1. The comparative period will be followed by a period where all subject will receive GammaCore® for 4 weeks.After the subject signed the Consent Form for participation the baseline (visit1) data will be collected. Subject will be informed how to complete the 2 week diary during the run-in period During the run-in period, all subjects will use stable SoC according to their individual prescriptions. The subject will record as CH attack regarding duration and frequency and the use of medication and oxygen.

Once subjects have finalized the run-in period, they are randomized to continue in 4 weeks comparative period. During this period, the control group continues with stable SoC and the active group is provided with a GammaCore® device for prophylactic and acute treatment in addition to the stable SoC Subjects stimulate 3 x 2 times daily as part of the prophylactic treatment regimen (cervical vagal nerve). Three 90 second stimulations are self-administered by the subject with 5 minutes between each stimulation on the right side of the neck.

This preventive stimulation regimen is performed:

* First Daily Treatment - within 1 hour of waking
* Second Daily Treatment - 7-10 hours following the first daily treatment

Acute CH attack:

* 3 x 90 second treatments consecutively at the onset of pain or symptoms. If the attack is not aborted within 15 minutes the subject should be informed to take SOC abortive medication.
* If an acute cluster headache attack is treated with the GammaCore® device, the subject will try to work within the preventive treatment window to avoid a preventive treatment in the 2-hour refractory period following the acute treatment.

A total of minimally 6 stimulations for the preventive part and as needed for the acute attacks. The active group also continues with the stable SoC during the entire 4 weeks period. Both groups record all CH attacks in the diary together with medication and oxygen use. All adverse events shall also be recorded in the diary.

The end of the 4 week comparative period marks the completion of the randomized part of the study, however all subjects are provided the option to continue to a 4 week GammaCore® treatment with the same stimulation parameter as during the 4 week randomization period. All subjects randomized to the SoC group will receive training.

During the entire study period, subjects are allowed to take rescue medication including oxygen inhalation for abortion of CH attacks. The amount and doses of the medication and oxygen are recorded in the diary.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form 2. Subjects between the age of 18-70, both genders 3. Subjects diagnosed with chronic cluster headache for at least 1 year, without remission periods or with remission periods lasting <1 month, in accordance with the ICHD-II classification criteria (2ndEd):

a. At least 5 attacks fulfilling the following criteria: i. Severe or very severe unilateral orbital, supraorbital and/or temporal pain lasting 15-180 minutes if untreated ii. Headache is accompanied by at least 1 of the following:

1. Ipsilateral conjunctival injection and/or lacrimation
2. Ipsilateral nasal congestion and/or rhinorrhea
3. Ipsilateral eyelid oedema
4. Ipsilateral forehead and facial sweating
5. Ipsilateral miosis and/or ptosis
6. A sense of restlessness or agitation iii. Attacks have a frequency from 1 every other day to 8 per day and are not attributed to another disorder iv. Attacks recur over > 1 year without remission periods or with remission periods lasting < 1 month.

4. Has minimum mean attack frequency of 4 CH attacks per week. 5. Is able to distinguish CH from other headaches (i.e. tension-type headaches).

6. Is capable of completing headache pain self-assessments. 7. Agrees to use the GammaCore® device as intended and follow all of the requirements of the study, including follow-up visit requirements.

8. Is willing to keep all concomitant medication stable during the entire study period.

9. Women of child-bearing potential must use 2 methods of contraceptive i.e. hormones and condom.

Exclusion Criteria:

1. Is currently taking CH prophylactic medication for indications other than CH which in the opinion of the clinician may interfere with the study
2. Has had a change in type or dosage of prophylactic headache medications < 1 month prior to enrollment
3. Has a history of intracranial or carotid aneurysm, intracranial hemorrhage, brain tumors or significant head trauma.
4. Has a lesion (including lymphadenopathy), dysaesthesia, previous surgery or abnormal anatomy at the GammaCore® treatment site.
5. Has other significant pain problem that might confound the study assessments in the opinion of the investigator.
6. Has known or suspected severe atherosclerotic cardiovascular disease, severe carotid artery disease (e.g. bruits or history of TIA or CVA), congestive heart failure (CHF), known severe coronary artery disease or recent myocardial infarction (within 5years).
7. Has had a previous unilateral or bilateral vagotomy.
8. Has uncontrolled high blood pressure.
9. Is currently implanted with an electrical and/or neurostimulator device, including but not limited to cardiac pacemaker or defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, or cochlear implant.
10. Has a history of carotid endarterectomy or vascular neck surgery on the right side.
11. Has been implanted with metal cervical spine hardware or has a metallic implant near the GammaCore® stimulation site.
12. Has a history, the last 12 month, of syncope.
13. Has a history, the last 12 month of seizures.
14. Has a known history or suspicion of substance abuse or addiction, or overuse of acute headache medication for headaches other than CH.
15. Has psychiatric or cognitive disorder and/or behavioral problems which in the opinion of the investigator may interfere with the study
16. In the opinion of the investigator the subject is incapable of operating the GammaCore® device as intended and performing the data collection procedures.
17. Is participating in any other therapeutic clinical investigation or has participated in a clinical trial in the preceding 30 days.
18. Woman who are pregnant or lactating.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2012-10; Primary Completion 2014-03 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charly Gaul, Dr med, Principal Investigator — Migräne- und Kopfschmerzklinik Königstein
Locations (10):
- University Department of Neurology CHR, Liège, Liège, Belgium
- Germany (5):
  - Krankenhaus Lindenbrunn, Department of Neurology, Coppenbrügge, Coppenbrügge
  - Westdeutsches Kopfschmerzzentrum, Hufelandstr. 26, Hesse
  - Migräne- und Kopfschmerzklinik Königstein, Königstein im Taunus, Königstein Im Taunus
  - Department of Neurology, University of Munich, Munich, Munich
  - Neurologische Klinik und Poliklinik, Berlin, State of Berlin
- Regional Referral Headache Centre Sant' Andrea Hospital, Rome, Rome, Italy
- United Kingdom (3):
  - The Southern Hospital, Neurology Department, Glasgow, Scotland
  - Hull Royal Infirmary, Neurology Department, Hull
  - The Walton Centre, Neurology Department, Liverpool

IPD SHARING:
Plan to Share IPD: No
Not planned to share individual data

REFERENCES:
- [Derived] Morris J, Straube A, Diener HC, Ahmed F, Silver N, Walker S, Liebler E, Gaul C. Cost-effectiveness analysis of non-invasive vagus nerve stimulation for the treatment of chronic cluster headache. J Headache Pain. 2016;17:43. doi: 10.1186/s10194-016-0633-x. Epub 2016 Apr 22. PMID 27102120

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | GammaCore
Started | 49 | 48
FAS Unmatched Data | 48 (1 patient protocol violation) | 45 (3 patients protocol violation)
FAS Matched Data | 42 | 32
Completed | 37 | 33
Not Completed | 12 | 15
Not completed — Protocol Violation | 1 | 3
Not completed — Did not complete the open label period | 11 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | GammaCore | Total
Number analyzed (Participants) | 49 | 48 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (11.0) | 45.4 (11.0) | 43.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 33 | 34 | 67
Region of Enrollment [Number; unit: participants]
  Belgium | 5 | 4 | 9
  Germany | 28 | 29 | 57
  United Kingdom | 13 | 11 | 24
  Italy | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: A Change in the Frequency of Cluster Headache Attacks Per Week
Description: The primary endpoint is the reduction in mean number of CH attacks per week. The number of CH attacks will be calculated as the sum of all attacks over the days in the run-in period and divided by the number of weeks, respectively for the last 14 days of treatment during the randomised phase. The reduction will then be the number of CH attacks during treatment period (last 14 days of the randomized treatment period) - number of CH attacks during run-in.
Time Frame: 4 weeks
Population: Full analysis set (FAS), matched group.
Measure: Mean (Standard Deviation); unit: CH attacks per week
Arm/Group | Standard of Care | GammaCore
Number analyzed (Participants) | 48 | 45
CH attacks per week | -2.0 (7.6) | -7.6 (6.4)

2. Secondary Outcome: Pain Relief of Headache Attacks
Description: The median pain during baseline (2 weeks) will be compared with the last 14 days of the treatment period Scale 0-4 0= no pain
  1. mild pain
  2. moderate pain
  3. severe pain
  4. very severe pain
Time Frame: baseline (2 weeks) and random period(last 2 weeks)
Population: Median severity per subject in run in period (14 days) and the last 14 Days in the treatment period.
  FAS matched data set
Measure: Number; unit: participants
Arm/Group | Standard of Care | GammaCore
Number analyzed (Participants) | 42 | 32
participants
  Mild baseline | 2 | 1
  Mild random | 3 | 1
  Moderate baseline | 16 | 8
  Moderate random | 15 | 11
  Severe baseline | 16 | 15
  Severe random | 16 | 12
  Very severe baseline | 8 | 8
  Very severe random | 8 | 8

3. Secondary Outcome: Adverse Events
Description: The frequency of device effects will be compared between the two treatment groups. Only effects which are new after baseline or have increased severity after baseline will be used in the comparison.
Time Frame: 10 weeks
Population: Safety population The Adverse Device effects are reported as Adverse Event, the device effects are AEs that are considered related to the treatment. Graded mild, moderate and severe
Measure: Number; unit: participants
Arm/Group | Standard of Care | GammaCore
Number analyzed (Participants) | 49 | 48
participants
  Mild | 6 | 9
  Moderate | 2 | 1
  Severe | 0 | 1

4. Secondary Outcome: EQ-5D-3L (EuroQoL 5 Questions and 3 Answering Levels) and a VAS (Visual Analogue Scale)
Description: The EQ-5D-3L (EuroQoL 5 questions and 3 answering levels) during the run-in period will be compared with the EQ-5D-3L during the treatment period. And treatment period will be compared to open label.
  Rating of questions Level 1 no problems Level 2 some problems Level 3 Significant problems Worst case is 15 points and best case is 5 points using index
  Visual analogue scale VAS 0-100 where 0 is the worst imaginable health state and 100 the best imaginable health state
Time Frame: 10 weeks (baseline 2 weeks, random 4 weeks and open label 4 weeks)
Population: Changes between baseline and randomized period.Randomized period and open label. FAS Unmatched data.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Standard of Care | GammaCore
Number analyzed (Participants) | 48 | 45
units on a scale
  Baseline vs. Randomized period | -0.049 [-0.837 to 0.856] | 0.145 [-0.532 to 0.807]
  Randomized period vs. Open label perios | 0.078 [-0.601 to 1.01] | 0.155 [-0.568 to 1.01]
  VAS Baseline vs. Randomized period | 0.27 [-81.0 to 40.0] | 9.20 [-20.0 to 40.0]
  VAS Randomized period vs. Open label | 4.36 [-50.0 to 48.0] | 10.79 [-26.0 to 55.0]

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Standard of Care | GammaCore
Serious Adverse Events (participants affected / at risk) | 2/49 | 2/48
Other Adverse Events (participants affected / at risk) | 3/49 | 3/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=49) | GammaCore (N=48)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) — Hospitalization/Not related
Scrotal Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Hospitalization/Not related
Genital herpes simplex (Infections and infestations) | 1 (1) | 0 (0) — Hospitalization/Not related
Cluster headache (Nervous system disorders) | 1 (1) | 0 (0) — Hospitalization/Not related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=49) | GammaCore (N=48)
Dizziness (Nervous system disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No